CLINICAL TRIAL: NCT03994536
Title: Effectiveness of a Person-Centred Transition Program to Empower Adolescents With Type 1 Diabetes in the Transition to Adulthood: the STEPSTONES-DIAB Project
Brief Title: Effectiveness of a Transition Program for Adolescents With Type 1 Diabetes in the Transition to Adulthood
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Karolinska University Hospital (Other); Swedish Child Diabetes Foundation (Other); Swedish Diabetes Foundation (Unknown); Gothenburg Centre for Person-Centred Care (Unknown); The Swedish Research Council (Other Government); Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/1725-31
Record Dates: First submitted 2019-06-09; First posted 2019-06-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
Keywords: Transfer to adult care; Continuity of patient care; Transition program; Empowerment; Adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Empowerment | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: transition program (Experimental): Participants come from two clinics and will be randomly allocated to this group. Participants will go through a transition program which will last for 2 years. The intervention will be performed by specialist nurses (transition coordinators) who meet the participants at three occasions during the study period and participants will be offered to meet peers with type 1 diabetes during an adolescent day.
  Interventions: Behavioral: A Person-Centred Transition Program to Empower Adolescents With Type 1 Diabetes in the Transition to Adulthood: the STEPSTONES-DIAB Project
- Comparison group: Standard care (Experimental): Participants allocated to this group will receive usual care, which includes regular follow-up visits in pediatric diabetes outpatient clinics. Usual care can vary across the two clinics, however, they all include meetings with a nurse and a physician.
  Interventions: Other: Standard care

INTERVENTIONS:
Behavioral: A Person-Centred Transition Program to Empower Adolescents With Type 1 Diabetes in the Transition to Adulthood: the STEPSTONES-DIAB Project — Behavioral: Transition program Participants will be part of a transition program that aim to prepare them for adult life and adult care wich includes eight key components: 1. A transition coordinator; 2. Education on diabetes, treatments, health behavior, dealing with school, friends; 3. Telephone availability; 4. Information about the adult diabetes service: 5. Guidance of parents; 6. Meeting with peers: 7. A person-centered transition plan; and 8. Preparation and transfer to adult diabetes service.
  Arms: Intervention group: transition program
Other: Standard care — Participants allocated to this group will receive usual care, which includes regular follow-up visits in pediatric diabetes outpatient clinics. Usual care can vary across the two clinics, however, they all include meetings with a nurse and a physician.
  Arms: Comparison group: Standard care

SUMMARY:
The transfer of young people with type 1 diabetes (T1D) to adult care occurs during a critical period of life, while many young people with T1D have unsatisfactory glycemic control. The preparation to take over responsibility for their health and self-care as well as increasing their participation in care are important aspects for strengthening people's own ability, an important component of person-centered care. STEPSTONES-DIAB aims to evaluate the effectiveness of a person-centred transition program for adolescents with T1D to empower them to become active partners in their care. The study is conducted at two hospitals in Stockholm, Sweden where 140 patients will be randomized to either a structured, person-centered transition program over a 2.5 -year period or to usual care. Outcome measures is empowerment, participation and responsibility in care, health status, glycemic control as well as the participants' experiences of care during transfer.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is one of the most common chronic diseases in childhood. Each year, nearly 86 000 children around the world develop T1D. The annual mean incidence rates varies from 0.1-60/100000 with Sweden as one of the "top" incidence countries. Within diabetes care, most health care professionals agree that a lack of effective transfer from pediatric to adult care may contribute to insufficient continuity of health care and increased risk for adverse outcomes in young adults with T1D diabetes. In order to help the adolescent in the transitions to adulthood and adult care, transitions programs have been proposed as a complex intervention with the objective of maximizing lifelong functioning and potential through appropriate healthcare services. Therefore, research on transition and transfer, and on interventions that have the potential to improve both these clinical processes, is important.

Patient empowerment is recognized as an essential element of transition interventions. Through the promotion of patient empowerment the adolescents can become active partners in their care and have the knowledge and capacity to make decisions that affect their life and health status. The purpose of this study is to assess the effectiveness of a transition program for adolescents with type 1 diabetes within a randomized controlled trial. During the course of the study, participants will be part of a transition program or receive usual care before being transferred to adult care. The primary outcome is level of empowerment and secondary outcomes include health behavior as well as diabetes specific and transfer specific variables.

The investigators will assess the effectiveness of the transition program by comparing the level of empowerment (primary outcome) between the participants who received usual care and those who participated in the transition program. A higher level of empowerment from the group part of the intervention is expected. The economic evaluation entails an impact budget assessment and a cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Literate
* Swedish-speaking
* Diagnosed with type 1 diabetes (one year duration)
* Age: 16 years

Exclusion Criteria:

* Conditions affecting cognitive abilities
* If other diagnosis are present, type 1 diabetes must be the primary diagnosis

Ages: 16 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Level of empowerment | Endpoint after 2.5 years from baseline
  Gothenburg Young Persons Empowerment Scale (GYPES) will be used to assess the level of empowerment. This scale was developed by the researchers involved in this study and has been tested in a previous cross sectional study in order to determine its psychometric properties in adolescents with congenital heart disease and type 1 diabetes.The five subscales measure: (a) self-perceived level of understanding of their disease (knowledge and understanding); (b) the capacity patients have to handle their disease (personal control); (c) the effect their illness has on their lives and sense of self (identity); (d) the capacity to make decisions along with the healthcare professional (shared decision-making); and (e) the ability to share their experiences and help others who are going through a similar situation (enabling others). The total score ranges from 15 to 75 points, with a higher score reflecting a higher level of empowerment.

SECONDARY OUTCOMES:
Transition readiness | Endpoint after 2.5 years from baseline
  Readiness for transition questionnaire RTQ (adolescent version). These questionnaires examine two aspects. First, the overall transition readiness is assessed, using two items ranging from 1 to 4. The sum of these two items results in a score ranging from 2 to 8. Second, the frequency of adolescent responsibility and parental involvement are reported in 10 different health behaviours, on a ﬁve-point Likert scale. Each variable results in a total score ranging from 10 to 40, and higher scores indicate higher adolescent responsibility or parental involvement, respectively.
Transition readiness | Endpoint after 2.5 years from baseline
  Readiness for transition questionnaire RTQ (parent version). These questionnaires examine two aspects. First, the overall transition readiness is assessed, using two items ranging from 1 to 4. The sum of these two items results in a score ranging from 2 to 8. Second, the frequency of adolescent responsibility and parental involvement are reported in 10 different health behaviours, on a ﬁve-point Likert scale. Each variable results in a total score ranging from 10 to 40, and higher scores indicate higher adolescent responsibility or parental involvement, respectively.
Transition readiness | Change from baseline (16 year) to 18.5 year
  Readiness for transition questionnaire RTQ (adolescent version)
Transition readiness | Change from baseline (16 year) to 18.5 year
  Readiness for transition questionnaire RTQ (parent version)
Health behavior | Endpoint after 2.5 years from baseline
  Health Behaviour Scale. Health behaviours are measured with the Health Behavior Scale-CHD. Health behaviours are 'activities a person undertakes to maintain or improve health and prevent diseases'.30 This scale assesses alcohol consumption, tobacco use, dental care and physical activity. The scale has 15 items that help to calculate three summary risk scores: substance use (score 0-100), dental hygiene (score 0-100) and total health risk score (score 0-100). Higher risk scores represent unhealthier behaviours.
Health behavior | Change from baseline (16 year) to 18.5 year
  Health Behaviour Scale. Health behaviours are measured with the Health Behavior Scale-CHD. Health behaviours are 'activities a person undertakes to maintain or improve health and prevent diseases'.30 This scale assesses alcohol consumption, tobacco use, dental care and physical activity. The scale has 15 items that help to calculate three summary risk scores: substance use (score 0-100), dental hygiene (score 0-100) and total health risk score (score 0-100). Higher risk scores represent unhealthier behaviours.
General Quality of Life | Endpoint after 2.5 years from baseline
  DISABKIDS Chronic Generic Measure - DCGM-12 measure general quality of life and the level of distress caused by a chronic disease.The short-form of the DISABKIDS chronic generic module consists of 12 five-point Likert-scaled items assigned to the three domains: mental, social and physical. Higher scores represents better outcome.
Health Related Quality of Life | Endpoint after 2.5 years from baseline
  DISABKIDS Diabetes Module (DM) consists of 13 five-point Likert scaled items and has two scales, an Impact and a Treatment scale. The Impact scale describes emotional reactions of needing to control every day life, and to restrict one's diet, the Treatment scale refers to carrying equipment and planning treatment. Higher scores represents better outcome.
Diabetes Burden | Endpoint after 2.5 years from baseline
  Check your Health measures self-perceived physical and emotional health, social relationships, and general QoL on four vertical thermometer scales, ranging from 0 to 100, with 0 indicating low self-perceived health. Each scale indicates self-perceived health with diabetes and, on the same scale, self-perceived health without diabetes. The measured difference between self-perceived health with and without diabetes is defined as the burden of diabetes.
HbA1c | Endpoint after 2.5 years from baseline
  Glycaemic control measured as HbA1c (mmol/mol), using a capillary test and analysed using the DCA 2000 apparatus (Siemens Medical Solution Diagnostics, Mölndal, Sweden). Higher values represent av worse outcome.
HbA1c | Mean value during study period (16-18.5 year)
  Glycaemic control measured as HbA1c (mmol/mol), using a capillary test and analysed using the DCA 2000 apparatus (Siemens Medical Solution Diagnostics, Mölndal, Sweden). Higher values represent av worse outcome.
Hypoglycemic events | From baseline (16 year) to 18.5 year
  Number of severe hypoglycemic events requiring assistance from others. Higher numbers represent a worse outcome.
Diabetic ketoacidosis | From baseline (16 year) to 18.5 year
  Number of diabetic ketoacidoses requiring hospital care. Higher numbers represent a worse outcome.
Clinic attendance 1 | During and six month after study period
  Number of visits. Less number than recommended represent a worse outcome.
Clinic attendance 2 | Number of months between the last visit in pediatric care, pre-transfer and the first visit in adult care, post-transfer, assessed up to 2 years
  Time between last visit in pediatric care and first visit in adult care. Longer time between visits represents a worse outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Children's Outpatient Diabetes Clinics, Astrid Lindgrens Children's Hospital, Karolinska University Hospital, Stockholm, Huddinge
  - Children's Outpatient Diabetes Clinics, Astrid Lindgrens Children's Hospital, Karolinska University Hospital, Stockholm, Solna

IPD SHARING:
Plan to Share IPD: Yes
Coded files will be available only for research purposes. Information will be given after a letter with the intention of the study has been submitted to the Steering Committee who will determine whether to approve or deny the application.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Hilderson D, Moons P, Van der Elst K, Luyckx K, Wouters C, Westhovens R. The clinical impact of a brief transition programme for young people with juvenile idiopathic arthritis: results of the DON'T RETARD project. Rheumatology (Oxford). 2016 Jan;55(1):133-42. doi: 10.1093/rheumatology/kev284. Epub 2015 Aug 28. PMID 26320142
- [Background] Hilderson D, Westhovens R, Wouters C, Van der Elst K, Goossens E, Moons P. Rationale, design and baseline data of a mixed methods study examining the clinical impact of a brief transition programme for young people with juvenile idiopathic arthritis: the DON'T RETARD project. BMJ Open. 2013 Dec 2;3(12):e003591. doi: 10.1136/bmjopen-2013-003591. PMID 24302502
- [Background] Small N, Bower P, Chew-Graham CA, Whalley D, Protheroe J. Patient empowerment in long-term conditions: development and preliminary testing of a new measure. BMC Health Serv Res. 2013 Jul 8;13:263. doi: 10.1186/1472-6963-13-263. PMID 23835131
- [Background] Acuna Mora M, Sparud-Lundin C, Bratt EL, Moons P. Person-centred transition programme to empower adolescents with congenital heart disease in the transition to adulthood: a study protocol for a hybrid randomised controlled trial (STEPSTONES project). BMJ Open. 2017 Apr 17;7(4):e014593. doi: 10.1136/bmjopen-2016-014593. PMID 28420661
- [Background] Acuna Mora M, Sparud-Lundin C, Burstrom A, Hanseus K, Rydberg A, Moons P, Bratt EL. Patient empowerment and its correlates in young persons with congenital heart disease. Eur J Cardiovasc Nurs. 2019 Jun;18(5):389-398. doi: 10.1177/1474515119835434. Epub 2019 Mar 5. PMID 30834772
- [Background] Burstrom A, Acuna Mora M, Ojmyr-Joelsson M, Sparud-Lundin C, Rydberg A, Hanseus K, Frenckner B, Nisell M, Moons P, Bratt EL. Parental uncertainty about transferring their adolescent with congenital heart disease to adult care. J Adv Nurs. 2019 Feb;75(2):380-387. doi: 10.1111/jan.13852. Epub 2018 Oct 18. PMID 30209810
- [Background] Acuna Mora M, Luyckx K, Sparud-Lundin C, Peeters M, van Staa A, Sattoe J, Bratt EL, Moons P. Patient empowerment in young persons with chronic conditions: Psychometric properties of the Gothenburg Young Persons Empowerment Scale (GYPES). PLoS One. 2018 Jul 20;13(7):e0201007. doi: 10.1371/journal.pone.0201007. eCollection 2018. PMID 30028863
- [Derived] Brorsson AL, Bratt EL, Moons P, Ek A, Jelleryd E, Torbjornsdotter T, Sparud-Lundin C. Randomised controlled trial of a person-centred transition programme for adolescents with type 1 diabetes (STEPSTONES-DIAB): a study protocol. BMJ Open. 2020 Apr 14;10(4):e036496. doi: 10.1136/bmjopen-2019-036496. PMID 32295780